CLINICAL TRIAL: NCT05933473
Title: Clinical and Procedural Outcomes of Ostial Left Anterior Descending Artery Intervention With or Without Crossover to Left-main
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MA Abdelreheem, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Coronary interventions
Record Dates: First submitted 2023-04-07; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-LAD (Crossover stenting (CO)) (Active Comparator): Crossover stenting (CO) from the LM into the LAD, using standard provisional bifurcation techniques and proximal stent optimization (POT), where post dilatation was typically performed.
  Interventions: Procedure: Percutaneous coronary intervention
- ostial LAD (Ostial stenting(OS)) (Active Comparator): Ostial stenting of the LAD (OS) with no cross-over back to the LM.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — percutaneous intervention to oseal LAD with or without LM stenting

SUMMARY:
Prospective interventional study evaluating clinical and procedural outcomes of patients with ostial left anterior descending artery lesion PCI alone or crossover with left main artery

DETAILED DESCRIPTION:
Aim of the work:

1. Evaluate the clinical and procedural outcomes in patients undergoing percutaneous intervention (PCI) for ostial left anterior descending (LAD) lesions while comparing the outcomes between those treated with a stent crossing over (CO) to the left main (LM) versus ostial stenting (OS) alone.
2. Define predictors of success in Ostial LAD lesion PCI.

Patients and methods:

1)Patients:

Inclusion criteria:

1. Patients with Significant ostial LAD >50% stenosis within 5mm from ostium
2. Either chronic coronary syndrome (CCS) (ongoing symptoms despite medical therapy) or acute coronary syndrome (ACS) patients.
3. De-novo lesions.

Exclusion Criteria:

1. Those with coronary angiography results such as: (significant disease of the LM more than 40% or ostial left circumflex (LCX) greater than 50%).
2. Patients with protected LM.
3. In adherence to a dual antiplatelet regimen by enrolled patients within the first 12 months after the procedure.

Methods:

It is prospective cohort study on patients in Assiut university heart hospital catheterization lab. with ostial LAD lesion (median, 0.1.0) that will include baseline demographic, clinical, and angiographic data.

All patients will be thoroughly informed about the procedure's possible risks and benefits, as well as alternative therapeutic choices prior to the intervention, and obtained signed consent from all participants.

In all cases, percutaneous coronary interventions and stenting will be performed according to standard techniques either trans-radial or transfemoral approach.

All patients pre-treated with dual antiplatelet therapy, including aspirin and loading dose of either clopidogrel or ticagrelor.

Unfractionated heparin will be given to all patients during the procedure with a target activated clotting time of >250 seconds.

Two main strategies for treating ostial LAD lesions will be used and analyzed in this study:

1. Crossover stenting (CO) from the LM into the LAD, using standard provisional bifurcation techniques and proximal stent optimization (POT), where post dilatation was typically performed.
2. Ostial stenting of the LAD (OS) with no crossover back to the LM. The choice of the technique and the use of intravascular imaging (IVUS) depends on the discretion of the treating interventional cardiologist.

   * Patients included in our study will be subjected to:

     1. Detailed History.
     2. General and complete cardiac examination.
     3. 12-Leads ECG.
     4. Detailed Echocardiography. \ 5)Coronary angiography findings including:

A. Quantitative angiographic measurements:

1. Reference diameter (mm).
2. Diameter stenosis (%).
3. Lesion length and distance from LAD ostium(mm).
4. Medina classification.
5. Bifurcation angle.

B. Techniques used:

1. Ostial LAD stenting.
2. Crossover with LM. C. IVUS or angiography guided PCI.

Basic IVUS Measurement

The following basic measurements may be made with IVUS:

1. Minimum lumen diameter (MLD): the shortest diameter via lumen's center.
2. Minimum lumen area (MLA): the smallest area via the lumen's center.
3. Stenosis area: (reference lumen area - stenosis lumen area)/reference lumen area.
4. Plaque burden: (EEM area - lumen area) / EEM area .

D. Contrast volume (ml) E. Fluoroscopy time (min.) Data will be gathered during hospital admission and follow-up. In-hospital mortality and morbidity will be documented.

Follow up:

During the hospital admission:

Both techniques used by our operators in these cases will be overviewed and evaluated as regarding:

1. Angiographic success in target vessel defined as (residual stenosis ≤ 30% and TIMI flow grade 3) and side branch (SB) angiographic success (residual stenosis ≤ 50% and TIMI flow grade 3).
2. Procedural Success A successful PCI should achieve angiographic success without in-hospital major clinical complications (e.g., cardiac death, target vessel related MI, emergency coronary artery bypass surgery) during hospitalization
3. Clinical Success in the short term, a clinically successful PCI includes anatomic and procedural success with relief of signs and/or symptoms of myocardial ischemia after the patient recovers from the procedure.

Information about the in-hospital outcome will be obtained from an electronic clinical database for patients maintained at our institution and by review of hospital records for those discharged to referring hospitals.

Short term follow up (after 6 months):

1. Per our institutional protocol, clinical follow-up will be performed by physicians in outpatient clinic after 4 months.
2. Control coronary angiography will be scheduled at 6 months to all cases.
3. Information on the occurrence of cardiac death, target vessel related myocardial infarction or repeated revascularization during period of follow-up will be collected by consulting our institutional electronic database and by contacting referring physicians and institutions and all living patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Significant ostial LAD >50% stenosis within 5mm from ostium
2. Either CCS (ongoing symptoms despite medical therapy) or ACS patients.
3. De-novo lesions.

Exclusion Criteria:

1. Those with coronary angiography results such as: (significant disease of the LM more than 40% or ostial LCX greater than 50%).
2. Patients with protected LM.
3. In adherence to a dual antiplatelet regimen by enrolled patients within the first 12 months after the procedure.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the clinical outcomes using different techniques in ostial LAD | 6 months
  Evaluate the clinical outcomes in patients undergoing PCI for ostial LAD lesions
  The primary end points are:
  -Target vessel related myocardial infarction occuring within 48 hours defined by absolute rise in cardiac troponin (from baseline) ≥35 times upper reference limit plus 1 (or more) of the following criteria:
  * Flow-limiting angiographic complications.
  * New "substantial" loss of myocardium on imaging.

SECONDARY OUTCOMES:
Predictors of PCI success | 6 months
  -Angiographic success in target vessel defined as residual stenosis ≤ 30% and TIMI flow grade 3
Predictors of PCI success | 6 months
  -Angiographic success in target vessel defined as SB angiographic success (residual stenosis ≤ 50% and TIMI flow grade 3).
Predictors of ostial LAD PCI success | 6 months
  -Procedural Success by doing successful PCI without in-hospital major clinical complications wihin one week of hospitalizaion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AN AbdEl-Reheem, MSC, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Background] Rigatelli G, Zuin M, Baracca E, Galasso P, Carraro M, Mazza A, Lanza D, Roncon L, Daggubati R. Long-Term Clinical Outcomes of Isolated Ostial Left Anterior Descending Disease Treatment: Ostial Stenting Versus Left Main Cross-Over Stenting. Cardiovasc Revasc Med. 2019 Dec;20(12):1058-1062. doi: 10.1016/j.carrev.2019.01.030. Epub 2019 Jan 31. PMID 30797760
- [Background] Guidelines for percutaneous transluminal coronary angioplasty. A report of the American College of Cardiology/American Heart Association Task Force on Assessment of Diagnostic and Therapeutic Cardiovascular Procedures (Committee on Percutaneous Transluminal Coronary Angioplasty). J Am Coll Cardiol. 1993 Dec;22(7):2033-54. No abstract available. PMID 8245363
- [Background] Frangos C, Noble S, Piazza N, Asgar A, Fortier A, Ly QH, Bonan R. Impact of bifurcation lesions on angiographic characteristics and procedural success in primary percutaneous coronary intervention for ST-segment elevation myocardial infarction. Arch Cardiovasc Dis. 2011 Apr;104(4):234-41. doi: 10.1016/j.acvd.2011.02.001. Epub 2011 Apr 19. PMID 21624790